CLINICAL TRIAL: NCT07194863
Title: Efficacy of Essential Phospholipid Versus Betaine HCL/L-Glutamic Acid in MAFLD
Acronym: EssenMAFLD
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Mohammed Abdel Mowgod, Efficacy of Essential phospholipid versus Betaine HCL/L-Glutamic Acid in MAFLD, Assiut University
Other Study IDs: 2025-04-300571
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-09

CONDITIONS: Essential Phospholipid in Metabolic Associated Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * After obtaining the appropriate consents, data pertaining to clinical history (name, age, sex, residence, occupation, co-morbidities… diabetes, hyperlipidemia, hypertension, ischemic heart disease, special habits; such as alcohol intake).
  * Imaging techniques, such as ultrasonography (US), fibroscan with CAP and/or computed topography (CT) and /or MRI.
  * Blood samples will be collected for liver function tests (albumin, alanine aminotransferase [ALT], aspartate aminotransferase [AST], blood sugar, gamma-glutamyl transpeptidase, total bilirubin), lipid profile (total cholesterol, triglyceride, LDL) and CRP.
  * Six measurements will be obtained (sex, age, height, weight, body mass index, and abdominal girth, waist circumference). Calculation of fatty liver index, (FLI) will be done. The fatty liver index (FLI), is an algorithm based on waist circumference, body mass index (BMI), triglyceride, and gamma-glutamyl-transferase (GGT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the efficacy of Essential phospholipid versus Betaine HCL/L-Glutamic Acid in MAFLD

DETAILED DESCRIPTION:
The prevalence of non-alcoholic fatty liver disease (NAFLD) increases rapidly in recent decades. NAFLD has become a major public health problem in the whole world, and it is considered as the main cause for the chronic liver diseases (Egyptian study was done and recently published an international expert consensus statement about a new definition of metabolic dysfunction-associated fatty liver disease (MAFLD) to replace non-alcoholic fatty liver disease (NAFLD). The new nomenclature of MAFLD is based on the presence of steatosis in >5% of hepatocytes and the absence of excessive alcohol consumption or other causes of chronic liver disease, diagnosis of MAFLD could be established on the presence of hepatic steatosis in combination with one of the following three criteria: overweight/obesity; presence of type 2 diabetes mellitus; or evidence of metabolic dysregulation . Metabolic dysregulation is defined as having at least 2 of the following metabolic risk abnormalities: high waist circumference, high blood pressure, high cholesterol, pre-diabetes, insulin resistance, and high plasma C-reactive protein levels (2).New diagnostic criteria for MAFLD were proposed, in which hepatic steatosis (HS) detected either by imaging techniques, blood biomarkers/scores or by liver histology.On the other hand, NAFLD is commonly associated with one or more component of metabolic syndrome such as obesity, diabetes mellitus, and dyslipidemia and is defined as the presence of ≥ 5% hepatic steatosis in histological examination without evidence of hepatocellular injury such as hepatocyte ballooning (5).Around 20% of patients with NAFLD develop non-alcoholic steatohepatitis (NASH) which may progress to cirrhosis, however the most common cause of death in NAFLD patients is cardiovascular disease, and NAFLD is the third most common cause of hepatocellular carcinoma.The spectrum of NAFLD ranges from simple fatty liver with little inflammation to non-alcoholic steatohepatitis (NASH) with liver inflammation and fibrosis. The global prevalence of NAFLD is about 25.2% whereas the limited number of studies from Africa reports 13%."Burned out" NAFLD can be a hidden cause of cryptogenic cirrhosis. So, early diagnosis, and treatment of NAFLD and underlying predisposing factors are important to avoid liver damage which may progress to liver cell failure. NAFLD is strongly associated with MS and is currently considered as the hepatic manifestation of MS. In addition, obesity is a common risk factor for NAFLD. Essential phospholipids (EPLs) are naturally occurring hepatoprotective agents that have been used in the management of NAFLD. EPLs are obtained from soybeans, and their main component is phosphatidylcholine. EPLs improved liver steatosis in patients with NAFLD in a number of randomized controlled clinical trials, including placebo-controlled studies. The Russian guidelines for the diagnosis and management of NAFLD recommend EPLs as an adjunctive therapy for the management of NAFLD.

Subjective self-assessed parameters are measured in observational studies, usually without objective endpoints. NAFLD is almost always asymptomatic, so it is interesting that subjective feelings are a reliable indicator of objective disease severity. EPLs have been associated with subjective improvements, treatment satisfaction, and high adherence ; however, to date, no studies have analyzed whether subjective improvement, satisfaction with treatment, and adherence to treatment are associated with objective changes in liver structure or function. Mitochondrial dysfunction increases DNA methylation, which can cause the development of metabolic syndrome in obesity and the progression of NAFLD. Therefore, the regulation of DNA methylation could prevent NAFLD by attenuating mitochondrial dysfunction. DNA cytosine-5-methyltransferases (DNMTs) mediate DNA methylation by catalysing the transfer of the methyl group from SAM to cytosine during DNA replication. Betaine supplementation significantly elevates DNMT at the mRNA level in animals. The epigenetic effects of SAM via DNA methylation are driven by SAM precursors such as betaine and Met. Betaine acts as a methyl donor for DNA methylation in epigenetic regulation and provides a methyl group to participatein one-carbon metabolism to promote SAM formation. Recent research reported that access to 1% betaine-supplemented water for a total of 8 weeks alters the methylation status of specific gene promoters in mice, leading to persistent changes in gene expression that could be beneficial for the treatment of obesity and type 2 diabetes owing to their valuable metabolic effects on lipolysis, the TCA cycle and mitochondrial oxidative demethylation. However, the mechanism by which betaine methylation regulates mitochondrial oxidative demethylation to ameliorate NAFLD remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged >18 years old
* diagnosed as fatty liver based on clinical examination, laboratory investigations and imaging techniques.

Exclusion Criteria:

* Patients aged ≤18 years old.
* Pregnancy.
* Presence of malignancy.
* Type I DM.
* Fatty liver patients on treatment by statin derivatives or other medications.
* Fatty liver patients undergone bariatric surgeries

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * After obtaining the appropriate consents, data pertaining to clinical history (name, age, sex, residence, occupation, co-morbidities… diabetes, hyperlipidemia, hypertension, ischemic heart disease, special habits; such as alcohol intake).
  * Imaging techniques, such as ultrasonography (US), fibroscan with CAP and/or computed topography (CT) and /or MRI.
  * Blood samples will be collected for liver function tests (albumin, alanine aminotransferase [ALT], aspartate aminotransferase [AST], blood sugar, gamma-glutamyl transpeptidase, total bilirubin), lipid profile (total cholesterol, triglyceride, LDL) and CRP.
  * Six measurements will be obtained (sex, age, height, weight, body mass index, and abdominal girth, waist circumference). Calculation of fatty liver index, (FLI) will be done. The fatty liver index (FLI), is an algorithm based on waist circumference, body mass index (BMI), triglyceride, and gamma-glutamyl-transferase (GGT). Score varies from zero to100.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
evaluate the efficacy of Essential phospholipid versus Betaine HCL/L-Glutamic Acid in MAFLD | Baseline and at 12 weeks of treatment
  Evaluation of the mean change in hepatic fat fraction from baseline to the end of treatment to compare the efficacy of Essential phospholipid versus Betaine HCL/L-Glutamic Acid in patients with metabolic dysfunction-associated fatty liver disease (MAFLD).